CLINICAL TRIAL: NCT04194567
Title: An Absorption Study in Young Women to Evaluate the Effect of Polyphenols on Iron Absorption From Ragi (Finger Millet) Using the Iron Isotopic Method
Brief Title: Effect of Polyphenols on Iron Absorption From Finger Millet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Ragi
Record Dates: First submitted 2019-11-21; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Iron-deficiency
Keywords: polyphenols; iron deficiency; finger millet; iron bioavailability
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: The study will have a randomized, cross-over design and will be conducted at the Human Nutrition Laboratory, ETH Zurich (scientific responsibility). From an initial screening of 150 women, 25 non-pregnant non-lactating women with a marginal iron status (PF <25 ng/ml) will be recruited. In total, participants will consume the 2 intervention products in a random, balanced order. Participants will consume the first intervention product as a breakfast meal for 5 days in a week, and the second intervention product as a breakfast meal as well for 5 days the following week. A blood sample will be collected 14 days after the last meal administration day which will be used to measure the shift in the isotopic ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Ragi (Experimental): During one week of the study, participants are to consume pancakes made from the dark variety of ragi.
  Interventions: Other: Black Ragi
- White Ragi (Experimental): During the second week of the study, participants are to consume pancakes made from the white variety of ragi
  Interventions: Other: White Ragi

INTERVENTIONS:
Other: Black Ragi — Pancakes made out of the dark ragi
  Arms: Black Ragi
Other: White Ragi — Pancakes made out of the white ragi
  Arms: White Ragi

SUMMARY:
In India, one of the fast growing countries, 53% of all women have anaemia as per the National Family Health Survey. A recently published study on the burden of disease in India concluded that the burden of Iron deficiency anaemia (IDA) is 3 times higher than the average globally for other geographies at a similar level of development, and that women are disproportionately affected. Finger Millet (Eleusine coracana), more commonly known as Ragi, is a type of a millet crop grown in India, is considerably rich in minerals and its micronutrient density is higher than that of the world's major cereal grains: rice and wheat. Ragi also contains different antinutrients such as phytates and polyphenols, which have been known to have an inhibiting effect on the absorption of iron. On an average, white finger millet contains 0.04-0.09% polyphenols and brown varieties have 0.08-3.47%. The dark variety of ragi is the most widely consumed type. The white ragi is the lesser consumed type. However, the levels of polyphenols, which inhibit the absorption of iron, are ten times lower in the white ragi as compared to the dark ragi. Thus, it is important to evaluate the extent of inhibition of the polyphenols on the iron absorption. This information would be beneficial for policy making and promotion of cultivation of the type of ragi that could be most effective for the consumers

DETAILED DESCRIPTION:
Finger Millet (Eleusine coracana), more commonly known as Ragi, is a type of a millet crop grown in India, including other countries especially in East Africa. Ragi has been perceived as a potential "super cereal" by the United States National Academies being one of the most nutritious among all major cereals. From the nutritional perspective, finger millet is considerably rich in minerals and its micronutrient density is higher than that of the world's major cereal grains: rice and wheat .

Millets (Ragi or finger millet and Jowar or sorghum) were consumed by 59% of rural and 28% of urban population in Karnataka. Ragi consumption was seen predominantly in south Karnataka with 27% of rural and 17% of urban population reporting consumption.

Ragi is the richest source of calcium among cereals with up to 10-fold higher calcium content than brown rice, wheat or maize and three times than that of milk. It is also rich in iron and fiber, making this crop more nutritive as compared to other most commonly used cereals. Finger millet is enriched in the essential amino acids like lysine and methionine which are important in human health and growth but remain absent from most other plant foods . In addition, it also contains useful amounts of the two polyunsaturated fatty acids- linoleic acid and α-linolenic acid , metabolized products of which facilitate normal development of the central nervous system. Despite the well-documented health benefits of finger millet, only a limited progress has been made in context to its nutraceutical applications as functional food. Although, it may have remained underutilized by the general population due to either unawareness or apprehension, its immense potential for enhancing the nutritional and therapeutic attributes by acting as functional food cannot be ignored.

Ragi also contains different antinutrients such as phytates and polyphenols, which have been known to have an inhibiting effect on the absorption of iron. On an average, white finger millet contains 0.04-0.09% polyphenols and brown varieties have 0.08-3.47% . It was found that found proto-catechuic acid (45.0 mg/100 g) is the major free phenolic acid in ragi. In another study of total phenolic compounds in finger millet, it was found to have 85% benzoic acid derivatives (gallic acid, protocatechuic acid, p-hydroxybenzoic acid, vanillic acid, syringic acid) while rest of the fraction were either cinnamic acid derivatives (ferulic acid, trans-cinnamic acid, p-coumaric acid, caffeic acid, sinapic acid) or flavonoids (quercetin, Proanthocyanidins like condensed tannins) . Among bound phenloic acids, ferulic and p-coumaric acid are the major fractions and account for 64-96 and 50-99% of total ferulic and p-coumaric acid content of finger millet grains, respectively.

The dark variety of ragi is the most widely consumed type. The white ragi is the lesser consumed type. However, the levels of polyphenols, which inhibit the absorption of iron, are ten times lower in the white ragi as compared to the dark ragi. Thus, it is important to evaluate the extent of inhibition of the polyphenols on the iron absorption. This information would be beneficial for policy making and promotion of cultivation of the type of ragi that could be most effective for the consumers

The study duration will be 26 days from the first day of the first meal administration till the last blood withdrawal . For each appointment, the participants will spend about 30 minutes at the Human Nutrition Laboratory at ETH Zurich, between 7 and 9 am for breakfast meal consisting of pancakes made out of the ragi. the white ragi meal and the black ragi meal will be extrinsically labelled with isotopes 57 Fe and 58 Fe respectively. The participants will consume the ragi meal as breakfast. The first type of ragi meal will be given for 5 consecutive days,. They will have a weekend break of two days (during which they will resume their usual eating habits). After that, they will consume the second test meal as breakfast for another five consecutive days. Thus, there will be 10 meals in total. The breakfast meals will be consumed between 7 and 9 am together with a glass of 300 mL bottled water after which they have to wait another 3 hours before they can consume anything. The procedure will remain the same for all the days. Participants will always be asked to fast the day before coming for the feeding, that is, no food intake after 8 pm and no beverage intake after midnight the evening before. On day of screening, day 1 and the end point day 26 of the study, blood samples will be collected after an overnight fast for the determination of Hb, PF, CRP and isotopic ratio

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 40 years old
* Body weight up to 65 kg
* Normal Body Mass Index (18.5 - 25 kg/m2)
* Signed informed consent
* Plasma ferritin < 25 ng/ml
* Able to communicate in and comprehend English language
* Tasted and found the Ragi to be of acceptable taste and confirmed will to consume the test meals if enrolled in the study

Exclusion Criteria:

* Pregnancy (assessed by a urinary pregnancy test) / intention to become pregnant
* Lactating up to 6 weeks before study initiation
* Moderate or severe anaemia (Hb < 9.0 g/dL)
* Elevated CRP (> 5.0 mg/L)
* Any metabolic, gastrointestinal, kidney or chronic disease such as celiac disease, diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement)
* Continuous/long-term use of medication during the whole study (except for contraceptives)
* Consumption of mineral and vitamin supplements within 2 weeks prior to first meal administration
* Blood transfusion, blood donation or significant blood loss (accident, surgery) within 4 months prior to first meal administration
* Earlier participation in a study using iron stable isotopes or participation in any clinical study within the last 30 days
* Participant who cannot be expected to comply with study protocol (e.g. not available on certain study appointments or difficulties with blood withdrawal)
* Inability to understand the information sheet and the informed consent form due to cognitive or language reasons

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants enrolled in the study
Enrollment: 22 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Fractional Iron absorption | 26th day of the study
  The fractional iron absrption will be compared in predefined comparisons from the two interventions products that are administered to the study participants
Total Iron Absorption | 26th day of the study
  Total iron absorption from the two ragi types will be compared by measuring the total iron absorbed from all the meals in the study

SECONDARY OUTCOMES:
Hemoglobin | screening (-1), baseline (day 1), last test meal consumption (day 26)
  Iron status marker
Plasma ferritin | screening (-1), baseline (day 1), last test meal consumption (day 26)
  Iron status marker
C-Reactive Protein | screening (-1), baseline (day 1), last test meal consumption (day 26)
  Inflammation status
Body Iron stores | last test meal consumption (day 26)
  Iron status marker
Soluble transferrin receptor | last test meal consumption (day 26)
  Iron status marker

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - ETH Zürich, Laboratory of Human Nutrition, Zurich, Canton of Zurich
  - ETH Zurich, Laboratory of Human Nutrition, Zurich